CLINICAL TRIAL: NCT05787366
Title: Effect of a Health Pathway for People With Persistent Symptoms Covid-19
Acronym: SPACO+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22CH550; 2020-A00982-37 (Other: ANSM)
Record Dates: First submitted 2023-03-24; First posted 2023-03-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
Keywords: health pathway; quality of life; personalized multifactorial intervention
MeSH Terms: conditions — COVID-19 | interventions — Inosine Monophosphate

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, controlled, randomized open-labelled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Other): usual care and follow-up by a nurse: control group receiving conventional management, i.e. referral to a specialist(s) according to symptoms, as well as nursing follow-up.
  Interventions: Other: usual care and follow-up by a nurse
- Intervention group (Experimental): usual care and Personalized Multifactorial Intervention: group benefiting from the Personalized Multifactorial Intervention coordinated by a nurse
  Interventions: Other: Personalized Multifactorial Intervention (IMP)

INTERVENTIONS:
Other: usual care and follow-up by a nurse — follow-up by a nurse and referral to a specialist(s) according to symptoms
  Arms: Usual care
Other: Personalized Multifactorial Intervention (IMP) — The content of the intervention is defined according to the result of the initial assessment in relation to the person's needs and the nature of his or her persistent symptoms. The patient, depending on his or her needs, may choose to participate in the following workshops :
  * Knowledge of the disease and specific management, (led by the nurse)
  * Covid-19 and anxiety/depression, (psychologist)
  * Fatigue and adapted physical activities (video capsules)
  * Covid-long and social link (professional and voluntary activities...) (social worker and/or nurse)
  * The Recovery Café aims to provide a space for patients to listen to each other and share their experiences around themes related to the different dimensions of recovery: medical and psychological, economic, professional, social and existential.
  Arms: Intervention group

SUMMARY:
People with persistent symptoms of covid-19 have increased needs for needs for management of their overall health (physical, psychological and social). Persistent covid-19 symptoms have a negative impact on quality of life. By proposing a follow-up and an intervention on the reduction of these symptoms, the symptoms, the study will improve quality of life.

ELIGIBILITY:
Inclusion Criteria

* Persons who have been infected with Covid-19.
* Person with persistent clinical signs of Covid-19 for more than 12 weeks, referred by one of the partner structures of the project. The persistent signs of Covid-19 are: fatigue which can be severe, neurological disorders neurological disorders (cognitive, sensory, headaches), cardio-thoracic disorders (pain and chest tightness, tachycardia, dyspnea, cough) and disorders of smell and taste. Pain, digestive disorders and skin disorders are also common.
* Person who has agreed to participate and has given informed consent to participate in the study

Exclusion Criteria:

* Refused to participate in the study
* Person under legal protection
* Person with severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
the evolution of the quality of life | at the end of the 6-month follow-up
  measurement of quality of life at the end of the 6-month follow-up assess by the SF-36 questionnaire. This questionnaire has eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Each question is evaluated on a Likert scale, with 3, 5 or 6 levels of possible answers. The 8 dimensions are also used to calculate two quality of life scores for individuals: the physical composite score (PCS) and the mental composite score (MCS). The higher the score, the greater the ability.

SECONDARY OUTCOMES:
impact on quality of life | at 3 months
  Measuring the impact on quality of life assess by the SF-36 questionnaire. This questionnaire has eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Each question is evaluated on a Likert scale, with 3, 5 or 6 levels of possible answers. The 8 dimensions are also used to calculate two quality of life scores for individuals: the physical composite score (PCS) and the mental composite score (MCS). The higher the score, the greater the ability.
impact on frailty | at 3 and 6 months
  Measuring the impact on frailty by Fried frailty phenotype which assess 5 dimensions : Denutrition, Fatigue, Muscle weakness, Slowing down, Low level of physical activity.
impact on comorbidities | at 3 and 6 months
  Measuring the impact on comorbidities by Charlson comorbidity index. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found.
impact on dyspnea symptoms | at 3 and 6 months
  Measuring the impact on dyspnea symptoms with The Medical Research Council modified dyspnea scale. It is used to subjectively grade the severity of dyspnea in patients with chronic obstructive pulmonary disease (ranged 0-4).The higher the stage, the more severe the dyspnea.
impact on hyperventilation symptoms | at 3 and 6 months
  Measuring the impact on hyperventilation symptoms with the Nijmegen score. It is a score with sixteen items ranked from 0 (never occurs) to 4 (occurs, very often). A score ≥ 23/64 is suggestive of hyperventilation.
impact on fatigue symptoms | at 3 and 6 months
  Measuring the impact on fatigue symptoms with the Chadler fatigue scale. This is a 11-item scale divided into two components that measures physical fatigue and mental fatigue. Respondents can give a score of 0 to 3 to indicate how each statement applies to them, from "less than usual" to "much more than usual. The scores for each item are then summed to produce an overall score (ranged 0 to 33). Higher the score is, higher the fatigue is.
impact on neuropathic pain symptoms | at 3 and 6 months
  Measuring the impact on neuropathic pain symptoms with the DN4 questionnaire. At the end of the questionnaire, add up the 'yes' answers giving a total score out of 10. If the patients score is greater than or equal to 4, the test indicates that the patient is likely to be suffering from neuropathic pain.
impact on cognitive impairment symptoms | at 3 and 6 months
  Measuring the impact on cognitive impairment symptoms with the Montreal Cognitive Assessment. A maximum score out of 30 points will thus be obtained. Smaller the score is, higher the cognitive impairment is.
impact on musculoskeletal disorders symptoms | at 3 and 6 months
  Measuring the impact on musculoskeletal disorders symptoms with Nordic style questionnaire. The Nordic questionnaire is made up of closed questions, and can be used as a self-questionnaire or an interview. The questionnaire was created to answer the following question: "Does an osteoarticular pathology exist in the given population and if so, which body region does it affect?". Based on this idea, the questionnaire includes a diagram of the human body seen from behind, divided into nine anatomical regions. The question "have you at any time during the last 12 months or 7 days had a problem (pain, discomfort, discomfort)?" is asked for each anatomical region.
impact on post-exertional malaise | at 3 and 6 months
  Measuring the impact on post-exertional malaise. It consist of 10 questions with a Likert scale. Each question is said to be positive when the two associated scores (severity and frequency) are ≥ 2. Active post-exertional malaise are said to be present when at least one of the 5 situations questioned is positive.
impact on anxiety and drepssion | at 3 and 6 months
  impact on anxiety and drepssion via the HAD questionnaire. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21)

OTHER OUTCOMES:
obstacles and levers to participation and adherence to the intervention, as well as the satisfaction of patients and professionals | at 3 and 6 months
  Evaluation of the obstacles and levers to participation and adherence to the intervention, as well as the satisfaction of patients and professionals via semi-directive interviews conducted by a sociologist during the implementation of the intervention
Effectivness of the intervention | at 6 months
  Assess the effectivness of the system through a cost-utility analysis

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ROCHE, PhD, Principal Investigator — CHU de Saint Etienne; Bienvenu BONGUE, phD, Study Director — Jean Monnet University
Locations (3):
- France (3):
  - Urps Medecins Libéraux Auvergne-Rhône-Alpes, Lyon
  - Chu Saint-Etienne, Saint-Etienne
  - DAC Loire, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamdem OL, Dupre C, Heugno V, Baudot A, Essangui E, Blanquet M, Guercon N, Fanget M, Bayet S, Vericel MP, Oustric P, Mbama Biloa Y, Shikitele Lola E, Nekaa M, Debellis M, Stierlam F, Mbia RF, Tatsilong O, Assomo Ndemba P, Ngan WB, Ndobo V, Ayina Ayina C, Mekoulou J, Ndom Ebongue MS, Celarier T, Ruiz L, Regnier V, Bika C, Ngo Sack F, Ngondi JL, Barth N, Mandengue SH, Roche F, Botelho-Nevers E, Eboumbou Moukoko CE, Nguefeu Nkenfou C, Hupin D, Bongue B, Guyot J. SPACO+: a mixed methods protocol to assessing the effectiveness of an educative intervention in patients with Long Covid. BMC Infect Dis. 2025 Apr 29;25(1):623. doi: 10.1186/s12879-025-10992-6. PMID 40301772